CLINICAL TRIAL: NCT02431286
Title: Evaluation of Palonosetron and Palonosetron/Aprepitant in Post Operative Nausea and Vomiting Incidence in Oncological Patients
Brief Title: Palonosetron Associated to Aprepitant in Prophylaxis of PONV
Acronym: PONV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NP297/12; 2012/11298-8 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2015-01-31; First posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: nausea and vomiting, postoperative; emesis, postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant; Sodium Chloride; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant (Experimental): patient will receive aprepitant 80 mg per os one hour before surgery; palonosetron and dexamethasone will be intravenously administered during surgery
  Interventions: Drug: Aprepitant; Drug: Dexamethasone
- placebo (Placebo Comparator): patient will receive placebo per os one hour before surgery; palonosetron and dexamethasone will be intravenously administered during surgery
  Interventions: Drug: Placebo; Drug: Dexamethasone

INTERVENTIONS:
Drug: Aprepitant — aprepitant will be administered in preoperative period; intravenous palonosetron and dexamethasone will be administered intraoperatively
  Other Names: Emend
  Arms: Aprepitant
Drug: Placebo — Placebo will be administered in the preoperative period; intravenous palonosetron and dexamethasone will be administered intraoperatively
  Other Names: Saline
  Arms: placebo
Drug: Dexamethasone — Dexamethasone and plonosetron will be administered intraoperatively in both groups, durong surgery
  Other Names: Decadron

SUMMARY:
The objective of this study is to investigate if aprepitant in association with palonosetron and dexamethasone could reduce the incidence of PONV in high-risk patients for this symptom, undergoing cancer surgery mastectomies.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a common anesthetic complication that occurs in approximately 30% of the surgical population and can reach up to 70% in high risk patients for PONV. Advances have been made to prevent PONV, but the incidence is still high in certain groups of patients. In high risk patients, pharmacologic intervention should consist of multimodal therapy, targeting different mechanisms of action. The objective of this study is to investigate if aprepitant in association with palonosetron and dexamethasone could reduce the incidence of PONV in high-risk patients for this symptom, undergoing cancer surgery mastectomies. METHODS: this is a randomized and double blind clinical trial. Female high-risk patients for PONV(Apfel score 3 or 4) scheduled for mastectomy that agree with the study and signed the informed consent, are randomly distributed into one of two groups: Group A, aprepitant 80 mg per os one hour before the surgery and Group B will receive placebo by the same route one hour before surgery, in a blinded way. After induction of anesthesia, dexamethasone 4 mg and palonosetron 0,075mg are intravenously administered to all patients. After the end of the surgery, a patient-controlled analgesia (PCA) device will be intravenously inserted in all patients. In the postoperative period, patients will be evaluated for nausea, vomiting and pain intensity in the recovery room and after 24 hours

ELIGIBILITY:
Inclusion Criteria:

* patients submitted to breast cancer surgery
* non smokers

Exclusion Criteria:

* any contraindication to one of the drugs
* mental disease
* inability to understand the method or refusal to participate in the research

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative nausea and vomiting | 24 hours
  intensity of nausea

SECONDARY OUTCOMES:
postoperative pain measured by Verbal and descriptive scale | 24 hours
  pain intensity in the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hazem a Ashmawi, phD, Study Director — University of Sao Paulo
Locations (1):
- Angela Maria Sousa, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Moon HY, Baek CW, Choi GJ, Shin HY, Kang H, Jung YH, Woo YC, Kim JY, Park SG. Palonosetron and aprepitant for the prevention of postoperative nausea and vomiting in patients indicated for laparoscopic gynaecologic surgery: a double-blind randomised trial. BMC Anesthesiol. 2014 Aug 10;14:68. doi: 10.1186/1471-2253-14-68. eCollection 2014. PMID 25165427
- [Result] George E, Hornuss C, Apfel CC. Neurokinin-1 and novel serotonin antagonists for postoperative and postdischarge nausea and vomiting. Curr Opin Anaesthesiol. 2010 Dec;23(6):714-21. doi: 10.1097/ACO.0b013e32833f9f7b. PMID 20871394
- [Derived] Grigio TR, Sousa AM, Magalhaes GGN, Ashmawi HA, Vieira JE. Aprepitant plus palonosetron for the prevention of postoperative nausea and vomiting after breast cancer surgery: a double blind, randomized trial. Clinics (Sao Paulo). 2020;75:e1688. doi: 10.6061/clinics/2020/e1688. Epub 2020 Sep 2. PMID 32901672